CLINICAL TRIAL: NCT03865498
Title: Using Twitter to Enhance the Social Support of Hispanic and Black Dementia Caregivers
Brief Title: Twitter Based Social Support for Hispanic and Black Dementia Caregivers
Acronym: Tweet-S2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sunmoo Yoon, Associate Research Scientist, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAS3305; R01AG060929-01 (NIH)
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Loneliness; Emotional Stress
Keywords: Family Caregivers; Dementia
MeSH Terms: conditions — Stress, Psychological; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hispanic dementia caregivers (Experimental): De-identified followers of our Hispanic dementia caregiver Twitter network will receive messages from the network (Twitter for Hispanic caregivers' intervention).
  Interventions: Behavioral: Twitter for Hispanic caregivers
- African American dementia caregivers (Experimental): De-identified followers of our African American dementia caregiver Twitter network will receive messages from the network (Twitter for African American caregivers' intervention).
  Interventions: Behavioral: Twitter for African American caregivers

INTERVENTIONS:
Behavioral: Twitter for Hispanic caregivers — This group will be asked to follow and use (i.e., retweet, reply, like) our Hispanic Twitter network for social support
  Arms: Hispanic dementia caregivers
Behavioral: Twitter for African American caregivers — This group will be asked to follow and use (i.e., retweet, reply, like) our African American Twitter network for social support.
  Arms: African American dementia caregivers

SUMMARY:
The prevalence of dementia is higher in Hispanics and African Americans than non-Hispanic Whites. Moreover, dementia caregivers often experience loneliness as well decreased health status. The expansion of social media use among Hispanics and African Americans, particularly Twitter - a short message service - offers great promise for improving social support. This study aims to evaluate changes of discussion topics, sentiment and networking styles (i.e., number of followers) among anonymous followers of our two Twitter networks; the African American/Black dementia caregiver group and the Hispanic dementia caregiver group.

DETAILED DESCRIPTION:
The study will utilize Twitter networks to post a daily message for dementia caregivers for a year, and set up a monthly group chat.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Black or Hispanic, living in the U.S. including the U.S. territories
* a dementia caregiver with any duration, able to speak English or Spanish/bilingual
* must agree to terms of conditions of use and privacy policy and rules of one of the two dementia caregiver network (Hispanic @dcnh, Black @dcnaab), the Twitter user agreement of the terms of service, Twitter privacy policy and Twitter rules including intellectual property, violence, misconduct, abuse behavior, private information and spam and security
* use a smartphone or a feature phone (i.e., a cell phone with text messaging)

Exclusion Criteria:

* do not have de-identified Twitter account, children, not a dementia family caregiver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 966 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunmoo Yoon, PhD, Principal Investigator — Associate Research Scientist in the Department of Medicine
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on flyer distribution via community outreach offline (10 brain and Alzheimer's disease community events, community outreach) and online (Twitter advertisement, emails to 920+ community leaders) between January 2022 and June 2023. The first participant was enrolled on January 12, 2022, and the last was enrolled on June 14, 2023.
Groups:
- African American Family Members of Persons With Alzheimer's Disease and Related Dementias: Participants in the African American caregiving Twitter community received a multimedia Tweet message daily for 365 days and was asked to use (i.e., retweet, reply, like) our network community; Group message started on November 1, 2022 until October 31, 2023.
  Message ingredient: an evidence-based social support Tweet message tailored to African American family members of persons with ADRD [dosage: 1 group message, dosage form: video and text, frequency: 1 group message daily, administration duration: a short video 20-50 seconds, a group message length 280 characters reading time 3 seconds]
- Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias: Participants in the Hispanic caregiving Twitter community received a multimedia Tweet message daily for 365 days and was asked to use (i.e., retweet, reply, like) our network community; Group message started on November 1, 2022 until October 31, 2023.
  Message ingredient: an evidence-based social support Tweet message tailored to Hispanic family members of persons with ADRD [dosage: 1 group message, dosage form: video and text, frequency: 1 group message daily, administration duration: a short video 20-50 seconds, a group message length 280 characters reading time 3 seconds]
Period: Overall Study
Arm/Group | African American Family Members of Persons With Alzheimer's Disease and Related Dementias | Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias
Started | 506 | 460
Per Protocol 6m (186 Days) | 463 | 400
Per Protocol 9m (274 Days) | 435 | 352
Per Protocol 12m | 359 | 291
Completed | 367 | 312
Not Completed | 139 | 148
Not completed — Lack of Efficacy | 12 | 11
Not completed — Lost to Follow-up | 125 | 133
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- African American Family Members of Persons With Alzheimer's Disease and Related Dementias: African American caregiving Twitter community received a multimedia Tweet message daily for 365 days and was asked to use (i.e., retweet, reply, like) our network community; Group message started on November 1, 2022 until October 31, 2023.
  Ingredient: an evidence-based social support Tweet message tailored to African American family members of persons with ADRD [dosage: 1 group message, dosage form: video and text, frequency: 1 group message daily, administration duration: a short video 20-50 seconds, a group message length 280 characters reading time 3 seconds]
- Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias: Hispanic caregiving Twitter community received a multimedia Tweet message daily for 365 days and was asked to use (i.e., retweet, reply, like) our network community; Group message started on November 1, 2022 until October 31, 2023.
  Ingredient: an evidence-based social support Tweet message tailored to Hispanic family members of persons with ADRD [dosage: 1 group message, dosage form: video and text, frequency: 1 group message daily, administration duration: a short video 20-50 seconds, a group message length 280 characters reading time 3 seconds]
- Total: Total of all reporting groups
Arm/Group | African American Family Members of Persons With Alzheimer's Disease and Related Dementias | Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias | Total
Number analyzed (Participants) | 506 | 460 | 966
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (15.6) | 49.1 (15.6) | 47.9 (15.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 333 | 313 | 646
  Male | 172 | 145 | 317
  Prefer not to answer | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 247 | 460 | 707
  Not Hispanic or Latino | 255 | 0 | 255
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 18 | 18
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 399 | 57 | 456
  White | 0 | 63 | 63
  More than one race | 107 | 317 | 424
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 506 | 460 | 966
Number of participants who do not engage in Twitter activities [Count of Participants; unit: Participants] | 471 | 447 | 918
Emotional Valence Score [Mean (Standard Deviation); unit: score on a scale] — Emotional valence (macro level) detected from text data (e.g., "This is so helpful": emotion score +4; "I am sad": emotion score -6). Emotional valence score ranges from -10 to +10; -10 indicates negative valence and +10 indicates positive valence.
  score on a scale | 0.149 (1.054) | 0.073 (0.713) | 0.113 (0.908)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who do Not Engage in Twitter Activities
Description: Macro level: The number of participants who do not engage in Twitter activities (i.e., retweet, reply, like, post) within the Twitter network for dementia caregivers
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | African American Family Members of Persons With Alzheimer's Disease and Related Dementias | Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias
Number analyzed (Participants) | 506 | 460
Participants | 246 | 226
Statistical Analysis 1: Comparison: African American Family Members of Persons With Alzheimer's Disease and Related Dementias; Hypothesis: There will be significant pre/post-intervention differences in isolated macro-level network structures for African American dementia caregiver networks; Test type: Superiority; p < 0.0001, McNemar — McNemar's Chi-squared test (paired) with continuity correction to the test slightly more conservative; Odds Ratio (OR) = 7.029, 95% CI 2-sided [4.919 to 10.323]
Statistical Analysis 2: Comparison: Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias; Hypothesis: There will be significant pre/post-intervention differences in isolated macro-level network structures for Hispanic dementia caregiver networks; Test type: Superiority; p < 0.0001, McNemar — McNemar's Chi-squared test (paired) with continuity correction to the test slightly more conservative; Odds Ratio (OR) = 17.385, 95% CI 2-sided [9.963 to 33.157]
Statistical Analysis 3: Comparison: African American Family Members of Persons With Alzheimer's Disease and Related Dementias vs Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias; There will be no significant differences in isolated macro-level network structure from Tweets between Hispanic and African American dementia caregiver networks; Test type: Superiority; p = 0.924, Chi-squared, Corrected — Pearson's Chi-squared test with Yates' continuity correction; Odds Ratio (OR) = 1.021, 95% CI 2-sided [0.787 to 1.325]

2. Primary Outcome: Emotional Valence Score
Description: Emotional valence (macro level) detected from text data (e.g., "This is so helpful": emotion score +4; "I am sad": emotion score -6). Emotional valence score ranges from -10 to +10; -10 indicates negative valence and +10 indicates positive valence.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | African American Family Members of Persons With Alzheimer's Disease and Related Dementias | Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias
Number analyzed (Participants) | 506 | 460
score on a scale | 1.404 (2.412) | 1.483 (2.229)
Statistical Analysis 1: Comparison: African American Family Members of Persons With Alzheimer's Disease and Related Dementias; Hypothesis: There will be significant pre/post-intervention differences in emotional valence score detected from Tweets for African American dementia caregiver networks; Test type: Superiority — Pre-post mean difference; p < 0.0001, a paired t-test; Mean Difference (Final Values) = 0.628, 95% CI 2-sided [0.513 to 0.742]
Statistical Analysis 2: Comparison: Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias; Hypothesis: There will be significant pre/post-intervention differences in emotional valence score detected from Tweets for Hispanic dementia caregiver networks; Test type: Superiority — Pre-post mean difference; p < 0.0001, a paired t-test; Mean Difference (Final Values) = 1.410, 95% CI 2-sided [1.189 to 1.631]
Statistical Analysis 3: Comparison: African American Family Members of Persons With Alzheimer's Disease and Related Dementias vs Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias; There will be no significant differences in emotional valence score detected from Tweets between Hispanic and African American dementia caregiver networks; Test type: Superiority; p = 0.600, t-test, 2 sided; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [-0.186 to 0.107]

3. Secondary Outcome: Number of Auto-detected Small Groups
Description: Meso level: number of small group automatically detected based on Twitter activities (i.e., retweet); for example 0 means no small-group activity detected, 7 small groups mean seven distinct cliques/grouping activities detected where the users are communicating, supporting and responding within our Twitter network.
Time Frame: 12 months
Measure: Number; unit: Auto-detected Small Groups
Arm/Group | African American Family Members of Persons With Alzheimer's Disease and Related Dementias | Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias
Number analyzed (Participants) | 506 | 460
Auto-detected Small Groups
  Pre | 259 | 231
  Post | 262 | 239

4. Secondary Outcome: Percentage of Balanced Triads
Description: Micro level: % balanced communication triad, 2 or 3 people responding and communicating with equal or similar frequency; 0 reflects non-optimal communication indicating domination, avoidance or ignorance. 8 means there are 8% triads who maintain healthy communication.
Time Frame: 12 months
Population: Triad census: Counts of each triad type within a network are determined by analyzing all possible combinations of connections of 16 possible communication styles among three nodes (a triad) in each conversation.
Measure: Number; unit: percentage of balanced triads
Units Other Than Participants: Triads
Arm/Group | African American Family Members of Persons With Alzheimer's Disease and Related Dementias | Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias
Number analyzed (Participants) | 506 | 460
Number analyzed (Triads) | 6608580 | 4064785
percentage of balanced triads
  Pre | 0.00 | 0.00
  Post | 0.21 | 0.34

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | African American Family Members of Persons With Alzheimer's Disease and Related Dementias | Hispanic Family Members of Persons With Alzheimer's Disease and Related Dementias
All-Cause Mortality (participants affected / at risk) | 0/506 | 0/460
Serious Adverse Events (participants affected / at risk) | 0/506 | 0/460
Other Adverse Events (participants affected / at risk) | 0/506 | 0/460

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/98/NCT03865498/Prot_SAP_000.pdf